CLINICAL TRIAL: NCT05091008
Title: The Safety and Efficacy of Ledipasvir/Sofosbuvir in the Treatment of Chronic Hepatitis C Virus Infection in Naïve Children
Brief Title: Treatment of Chronic Hepatitis C Infection by Ledipasvir/Sofosbuvir in Naïve Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Noaman, Lecturer, Mansoura University Children Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MansouaUCH0322
Record Dates: First submitted 2021-09-24; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic hepatitis C; Egyptian children; Sofosbuvir; Ledipasvir
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HCV without co-morbidities (Active Comparator): Ledipasvir-Sofosbuvir fixed-dose combination one tablet (90 mg Ledipasvir, 400 mg Sofosbuvir), orally once daily at a fixed time with or without food for 12 weeks
  Interventions: Drug: Ledipasvir-Sofosbuvir 90 Mg-400 Mg Oral Tablet
- HCV with co-morbidities (Active Comparator): Ledipasvir-Sofosbuvir fixed-dose combination one tablet (90 mg Ledipasvir, 400 mg Sofosbuvir), orally once daily at a fixed time with or without food for 12 weeks
  Interventions: Drug: Ledipasvir-Sofosbuvir 90 Mg-400 Mg Oral Tablet

INTERVENTIONS:
Drug: Ledipasvir-Sofosbuvir 90 Mg-400 Mg Oral Tablet — proper history was taken. HCV genotyping was done revealed GT 4 in all included patients. Basic ECG and abdominal US were performed prior to treatment. Concomitant HBV infection was excluded by HBs Ag and anti-HBc antibody HIV screening was done prior to treatment. Basic investigations were done prior to therapy. All included patients received Ledipasvir-Sofosbuvir fixed-dose combination one tablet (90 mg Ledipasvir, 400 mg Sofosbuvir), orally once daily at a fixed time with or without food for 12 weeks. Regular visits were arranged at 4, 8, and 12 weeks with easy access to the pediatric hepatology unit and the treating physician if any urgent problem in between the visits. Every visit, laboratory investigations were checked. Adverse events (after excluding other possible causes) were reported for the safety profile of the drug. The efficacy of the drug, HCV-RNA was assessed by quantitative real-time PCR at 4 weeks and after the end of the treatment course (12 weeks)

SUMMARY:
Chronic hepatitis C virus (HCV) infection represents a crucial health problem in children that greatly influence their quality of life. Many efforts have been directed toward the investment of effective drugs with high safety profiles and with oral administration for better compliance. The development of a new direct-acting antiviral (DAA) made it possible to achieve these goals.

DETAILED DESCRIPTION:
The calculated sample size of the study was ....participants at 5% level of significance and 80 % power, using the following formula:

N= (Z1-α/2+Z1-β) 2 σ1* σ2 / δ 2 This study aims to evaluate the safety and efficacy of the combined Sofosbuvir/ Ledipasvir regimen given for 12 weeks in children aged 12-18 years or weighing at least 35 kg with HCV genotype 4 infections.

Patients will receive Ledipasvir-Sofosbuvir fixed-dose combination one tablet (90 mg Ledipasvir, 400 mg Sofosbuvir) taken orally once daily at a fixed time with or without food for 12 weeks. Visits will be arranged at 4, 8, and 12 weeks. Patients will have easy access to the pediatric hepatology unit and the treating physician if any urgent problem happens in between the visits.

The SPSS software version 24, SPSS was used for data processing

ELIGIBILITY:
* Inclusion Criteria:

  * Chronic HCV infection (≥ 6 months).
  * Weighing at least 35 kg.
  * Treatment-naïve children with chronic HCV infection without cirrhosis or with compensated cirrhosis.
  * Parent or legal guardian must provide written informed consent.
* Exclusion Criteria:

  * Patients with comorbidity of chronic medical illness (decompensated heart disease, severe renal impairment (GFR < 30) or ESRD, uncontrolled DM).
  * Concomitant HBV or HIV infection.
  * Medications (Amiodarone, beta-blockers).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of Ledipasvir-Sofosbuvir fixed-dose combination one tablet (90 mg Ledipasvir, 400 mg Sofosbuvir), in children with treatment-Naïve, chronic HCV infection, genotype 4. | at 4 weeks after discontinuation of therapy
  Proportion of patients with negative PCR
Evaluate the efficacy of Ledipasvir-Sofosbuvir fixed-dose combination one tablet (90 mg Ledipasvir, 400 mg Sofosbuvir), in children with treatment-Naïve, chronic HCV infection, genotype 4. | At 12 weeks after discontinuation of therapy
  Proportion of patients still with negative PCR

SECONDARY OUTCOMES:
Evaluate the safety of Ledipasvir-Sofosbuvir fixed-dose combination one tablet (90 mg Ledipasvir, 400 mg Sofosbuvir), in children with treatment-Naïve, chronic HCV infection, genotype 4. | At 4 weeks after discontinuation of therapy
  Assessment of possible adverse effects
Evaluate the safety of Ledipasvir-Sofosbuvir fixed-dose combination one tablet (90 mg Ledipasvir, 400 mg Sofosbuvir), in children with treatment-Naïve, chronic HCV infection, genotype 4. | At 12 weeks after discontinuation of therapy
  Assessment of possible new adverse effects not detected at 4 weeks after discontinuation of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Noaman, MD, Study Director — Lecturer
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, Egypt